CLINICAL TRIAL: NCT00458874
Title: Better Adherence to Therapeutic Lifestyle Change Efforts (BATTLE) Trial
Brief Title: Better Adherence to Therapeutic Lifestyle Change Efforts Trial
Acronym: BATTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU#06-12025
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Disease
Keywords: CV risk factors; subclinical atherosclerosis; lifestyle intervention; motivation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receive CIMT Results (R-CIMT) (Experimental): This group will receive visual feedback of their CIMT results on a weekly basis.
  Interventions: Behavioral: CIMT results
- Withhold CIMT Results (W-CIMT) (No Intervention): The W-CIMT group will not receive their CIMT results until the end of their study participation.

INTERVENTIONS:
Behavioral: CIMT results — Both groups will receive a weekly confidential packet of scripted materials (e.g. educational materials, class schedules, feedback from diet/exercise logs). The R-CIMT group will also receive an CIMT report which contains a copy of one of their own ultrasound scans, with a comparison "normal" scan. This report will also include the CIMT thickness, an interpretation that states their measurements are in the highest quartile for persons of their age and gender, and associated CVD risk. "Interpreting Your CIMT Results" tutorial will be included in the first weekly packet to educate subjects on the detection of atherosclerosis with carotid ultrasound. The CIMT results are withheld from the W-CIMT group until the end of their study participation along with the CIMT tutorial.
  Arms: Receive CIMT Results (R-CIMT)

SUMMARY:
The purpose of this study is to determine whether knowledge of abnormal results from a noninvasive test for detection of subclinical atherosclerosis (carotid intima media thickness [CIMT]), in addition to knowledge of cardiovascular disease (CVD) risk factors, enhances adherence to healthy lifestyle behaviors in comparison to only CVD risk factor knowledge. We believe that participants with CVD risk factors who have knowledge of their own CIMT test results showing significant subclinical atherosclerosis will demonstrate better adherence to therapeutic lifestyle change (TLC) than those subjects from whom the CIMT test information is withheld.

DETAILED DESCRIPTION:
The outcomes of subjects randomized to receive their CIMT information (R-CIMT Group) will be compared to a control condition of subjects randomized to have their CIMT information withheld (W-CIMT Group) until the completion of a lifestyle intervention that is common to both groups. The rationale for this intervention is based on the Health Belief Model theory that risk awareness prompts action for behavioral change. In particular, our aim is to study the impact of a subject's own CIMT results, and not the impact of generic educational material related to CIMT and CHD risk, on adherence to a lifestyle change program. Subjects will not know the hypothesis of this study because this knowledge could potentially impact their behavior during the intervention. Also, subjects will not be told that only half of them will receive their CIMT information before the lifestyle intervention, since subjects could potentially infer the study hypothesis from this knowledge. To answer the question of whether CIMT results would be a useful motivational tool for adherence to lifestyle change recommendations, there needs to be a comparison group that does not have their CIMT results. Subjects will be clearly told in the consent process results that they may not receive results of their clinical testing, including the CIMT results, until the end of their participation in this study. Randomization will occur after subjects successfully complete a "run-in" period during screening, which introduces the lifestyle intervention and teaches the proper use of the data collection tools. At the beginning of each week in the randomized phase of the study, subjects will receive a confidential packet of scripted materials. Packets will contain identical information (e.g. educational materials, class schedules, feedback from diet/exercise logs) except that the R-CIMT group will also receive a report that contains a copy of one of their own ultrasound scans, with a comparison picture of a normal scan. This report will also include the CIMT thickness in each artery and an interpretation that states that their measurements are in the highest quartile for persons of their age and gender. Attached to the report will be a tutorial ("Interpreting Your CIMT Results") to more fully educate participants on detection of atherosclerosis with carotid ultrasound. Both the CIMT results report and the tutorial specifically couple the presence of significant subclinical atherosclerosis with increased risk for cardiovascular morbidity and mortality. (Appendix D). If subjects from whom CIMT information is withheld request their CIMT results during the study, they will be told that those results will be made available to them at the end of their participation in the study, which is consistent with the information they were given in the consent process. At the end of the study, subjects who were randomized to receive their CIMT information will be asked to complete a quiz (Atherosclerosis and CIMT Knowledge Assessment) to determine their comprehension of the CIMT information that had been provided to them at randomization (Appendix D).

Lifestyle Intervention

All randomized subjects will participate in a 12-week lifestyle intervention program that will be introduced and observed in the "run-in" period during screening. This intervention will incorporate strategies that have proven benefit in reduction of CVD risk including aerobic exercise, Mediterranean-type diet, and ongoing contact with weekly, on-site group sessions for lifestyle change education and support integrating Transtheoretical Stages of Change and Social Cognitive learning theories.74-76 To minimize the potential of unblinding research staff to the randomization assignment of a large number of subjects, subjects will enter the next available block of 12-weekly group sessions regardless of randomization assignment. To minimize the potential of unblinding study subjects to the study hypothesis, all subjects will be instructed to refrain from discussing any personal medical or information contained in their weekly packet received during the group support sessions. Randomization assignment will be known only to statistician/data management team.

Aerobic Exercise Physical activity is a pillar of any lifestyle intervention program because it improves cardiorespiratory and muscular fitness and promotes improvement of CHD risk factors including obesity, diabetes, hypertension, and hyperlipidemia. Based on each subject's baseline fitness and safety issues, a physical activity program (with a goal of 180 minutes of aerobic exercise per week by the end of the study) will be prescribed by an exercise physiologist and tailored to individual choices from various types of moderate intensity activities. Exercise is recommended to occur on most days of the week and for at least 10 minutes per session within a defined target heart rate range. After the "run-in" period, exercise will be unsupervised but assessed with a heart rate monitoring device and self-monitoring logs.

Diet A Mediterranean-type diet with caloric goals based on each subject's weight will be prescribed by a registered dietician. The composition of the diet is structured to encourage consumption of plant-based, minimally processed, seasonal foods including fruits, vegetables, whole grains, legumes, nuts, fish and poultry in preference to red meat, low-fat dairy products, and limited amounts of beneficial unsaturated oils such as olive oil. The recommended diet will have a maximum of 35% of total calories from fat, a maximum of 7% of total calories from saturated fat, and a minimum of 15% of total calories from protein. Subjects will be instructed in meal planning and food preparation. Structured menus will be offered as an option. Review of self-monitoring logs by the dietician will guide individual feedback during the "run-in" period and in the weekly communication packets during the randomized period.

Group Support Weekly on-site sessions will be held to stimulate social support for the lifestyle intervention. A structured curriculum focusing on goal setting, problem solving, and stress reduction will be presented by a trained facilitator with opportunity for open discussion. To reinforce the diet plan, a group meal and periodic food preparation demonstrations also will occur during these sessions.

ELIGIBILITY:
Inclusion Criteria:

* Military healthcare beneficiary
* Willing to modify current diet and exercise habits
* Two or more of following CVD risk factors (hypertension, hyperlipidemia, family history, tobacco use, BMI >/= 25 kg/m2)
* Metabolic syndrome

Exclusion Criteria:

* Clinical CVD or conditions that limit safe participation
* Individuals who participation would interfere with conduct of trial
* No significant preclinical atherosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in lifestyle program adherence | Baseline, Week 12
  A composite index of adherence to the TLC intervention was selected as the primary outcome measure since the main goal of this study is to assess the impact of CIMT imaging knowledge on change in lifestyle behaviors.

SECONDARY OUTCOMES:
CVD risk factors | Baseline, 12 weeks
C-reactive protein | Baseline, Week 12
Anxiety | Baseline, Week 2, Week 12
Atherosclerosis and CIMT Knowledge | Week 12
  Knowledge test will be given to R-CIMT group only.
Adherence to each lifestyle change program component | Baseline, Week 12
  Adherence information will be collected on diet, exercise and attendance at weekly on-site sessions
Motivation | Baseline, Week 12
Self efficacy | Baseline, Week 12
  Nutrition and exercise self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Randolph Modlin, MD, Principal Investigator — Walter Reed Army Medical Center; Marina N Vernalis, DO, FACC, Study Director — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (1):
- Walter Reed National Military Medical Center / Integrative Cardiac Health Project (ICHP), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walizer EM, Vernalis MN, Modlin RE. Influence of CIMT as a motivator for health behavior change in a heart health program. Circulation 2014;129:AP126.
- [Result] Walizer EM, Vernalis MN, Modlin RE. Adherence to a lifestyle intervention program not improved by visual knowledge of carotid intima atherosclerosis. Circ Cardiovasc Qual Outcomes 2013;6:A43.
- [Result] Walizer E, Kashani M, Eliasson A, Vernalis M. Integrative Cardiac Health Project risk score improves cardiovascular risk assessment in women with subclinical atherosclerosis. J Cardiovasc Nurs 2011; 26(4):265A.